CLINICAL TRIAL: NCT06178341
Title: Randomized, Controlled Study to Evaluate the Effectiveness of the Kata® Inhalations-App in Reducing Critical and Non-critical Handling Errors and Improving Adherence to Prescribed Drug Inhalation Therapy and Asthma Control in Adult Patients With Asthma
Brief Title: Effects of the Kata® Inhalations-App on Inhaler Handling Errors, Adherence, and Asthma Control in Patients With Asthma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VisionHealth GmbH (Industry)
Collaborators: Thoraxklinik-Heidelberg gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asthma-KaRe
Record Dates: First submitted 2023-11-23; First posted 2023-12-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Asthma; Asthma control; Adherence; Inhalation technique; Inhaler; Digital therapeutics; Smartphone application
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Multicenter study in up to 15 study sites in Germany that follows a randomized, controlled, parallel-group, adaptive two-stage design.
Who Masked: Outcomes Assessor
Masking Description: The Investigator, the subjects and the data analyst will not be blinded. The persons evaluating the recordings of inhalation maneuvers will be blinded to study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Kata Inhalations-App with the following functions:
  1. Inhalation reminder
  2. Inhalation trainer
  3. Health parameter documentation
  4. Diary
  5. Audio and video recording of user's inhalation maneuvers
  6. Provision of study-specific questionnaires
  7. Reminder to fill out study-specific questionnaires
  Interventions: Device: Kata Inhalations-App
- Control (No Intervention): Messinstrument ("Measurement")-App. Smartphone application with the following functions:
  1. Audio and video recording of user's inhalation maneuvers
  2. Provision of study-specific questionnaires
  3. Reminder to fill out study-specific questionnaires
  Note: the Messinstrument-App does not provide any inhalation training, inhalation reminders, or feedback.

INTERVENTIONS:
Device: Kata Inhalations-App — The Kata Inhalations-App is a digital product that bears a CE mark. The application provides algorithms to run an inhalation trainer. The inhalation trainer shows patients how to improve their inhalation maneuver in a simple and understandable way. For this purpose, the signals from the camera and microphone of the patient's smartphone are used to evaluate the individual steps of the inhalation maneuver in real-time to provide automatic, personalized feedback. Additional functions of the Kata Inhalations-App include the possibility to document health parameters and to receive inhalation reminders.
  After set-up, subjects will use the application on their own as an add-on to their usual therapy for asthma. The total duration of application use will be 13 weeks, 1 week use of the Messinstrument ("Measurement")-App for all subjects (Baseline period), followed by 12 weeks use of the Kata Inhalations-App (intervention) or the Messinstrument-App (control).
  Arms: Intervention

SUMMARY:
The Kata® App is a digital therapy assistant for patients with asthma who need to inhale their therapy. Kata features inhalation trainers that shows patients in a simple and understandable way how to improve their inhalation maneuver so that the drug reaches the lungs efficiently. The Kata® App aims to reduce inhalation errors and ensures that inhaled drugs are used as approved and prescribed. Kata has different trainers for different inhalation devices. This study investigates the possible positive effects of the Kata® Inhalation App.

The main goal of the study is to:

1. investigate the effect of using the Kata® App on adherence for inhaled drugs in adult asthma patients. It consists of two parts: the correct use of the inhalers; and compliance with the therapy, or how much the patient follows the therapy plan as prescribed.
2. investigate the effect of using the Kata® App on asthma symptoms and asthma control, as measured by the Asthma Control Test (ACT) questionnaire.

In addition, asthma-related quality of life, lung function, and ease of use of the app will be assessed during the study.

This multicenter study follows a randomized, controlled, parallel-group, adaptive two-stage design. The study includes two different groups: an intervention and a control group. At the beginning of the study, each patient is randomly assigned to one of these two groups. The total duration of the study is 13 weeks: 1 baseline week and 12 intervention weeks. During the baseline week, the intervention and control group both use the app with limited functionality. Kata records their inhalations but does not provide inhalation training or feedback. This is to first assess how well patients are able to use their inhaler(s) without receiving support. After the first week, the intervention group starts using the app with full functionality for 12 weeks, which means that the app provides them with inhalation training and personalized feedback. The control group continues to use the app with limited functionality for 12 weeks, that means that they continue to use the app to record their inhalations but do not receive any inhalation training or feedback. This study will compare the patients in the intervention and control group, to find out the effect of using the Kata® inhalation app on the number of errors patients make when using their inhaler, therapy compliance, and health-related outcomes (asthma control, quality of life, and lung function).

ELIGIBILITY:
Inclusion Criteria

A subject is eligible to be included in the study only if all of the following criteria apply:

Age

1. At least 18 years of age at the time of signing the informed consent.

   Sex
2. Male or female.

   Type of Subject and Disease Characteristics
3. Sufficient knowledge of the German language as assessed by the Investigator.
4. Capability to use a smartphone comfortably in the opinion of the Investigator: the subject uses a smartphone on a regular basis, and makes use of smartphone applications (i.e., uses the smartphone for more than calling and sending text messages).
5. Established diagnosis of asthma.
6. Regular use (i.e., at least once daily) of at least 1 of the following devices: metered-dose inhalers (MDIs), Respimat, NEXThaler, Ellipta, Easyhaler, Breezhaler and Turbohaler.
7. Stable disease (i.e., no exacerbation and/or change in treatment regimen) within the last 4 weeks prior to screening.

   Informed Consent
8. Provision of written informed consent prior to any study specific procedure.

Exclusion Criteria

Subjects are excluded from the study if any of the following criteria apply:

Medical Conditions

1. History or evidence of any clinically relevant and/or major disease that, in the opinion of the Investigator, would constitute a risk when taking part in the study or interfere with the interpretation of data.
2. Confirmed SARS-CoV-2 infection at screening.

   Prior/Concomitant Therapy
3. Previous use of the Kata Inhalations-App.

   Prior/Concurrent Clinical Study Experience
4. Use of any investigational drug or participation in any clinical study within 30 days prior to the expected date of first application of study intervention.
5. Previous randomization in this study.

   Other Exclusions
6. Employee of VisionHealth, the study site, the Nuvisan Group, or other Contract Research Organization involved in the study.
7. Legal incapacity or limited legal capacity, or incarceration.
8. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the protocol requirements, instructions, and study-related restrictions.
9. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Change in the average number of handling errors per inhalation compared between the intervention and control group | Change in average number of handling errors per inhalation from baseline (study week 1) to the final intervention week (study week 13)
  Based on the recordings of the inhalation maneuvers from each data collection period, the inhaler handling and inhalation technique of each subject will be evaluated centrally by trained blinded personnel, based on the applicable German Airway League checklists for inhalation maneuvers (Checklisten Deutsche Atemwegsliga).
Change in Asthma Control Test (ACT) score compared between the intervention and control group | Change in ACT score from baseline (study week 1) to the final intervention week (study week 13)
  The ACT consists of 5 questions (items) to assess the subject's asthma symptom control within the last 4 weeks. Each question can be answered on a 5-point numerical scale from 1 (worst) to 5 (best). The ACT score is the total score of all items. An ACT score of ≤ 15 points means "no asthma control", a score of 16 to 19 points means "partial asthma control" and a score of ≥ 20 points means "complete asthma control". These are the 3 ACT asthma control classes. The minimal clinically important difference for the ACT is 3 points.
  The ACT will be completed during each data collection period. The questionnaire will be made available within the smartphone application. Subjects will be reminded to complete the ACT.

SECONDARY OUTCOMES:
Change in the Test of Adherence for Inhalers (TAI) score (patient domain) compared between the intervention and control group | Change in TAI score from baseline (study week 1) to the final intervention week (study week 13)
  The TAI consists of 12 questions (items) to assess a subject's observance of inhalation therapy. The questions are grouped into 2 parts (domains) that can be scored and evaluated separately. In the 'patient domain', 10 items can be rated on a 5-point numerical scale from 1 (worst rating) to 5 (best rating). Based on the total score from those 10 questions, the extent of therapy observance (TAI adherence class) can be assessed: 50 points: adherent patients; 46 to 49 points: moderately adherent patients; ≤ 45 points: non-adherent patients. In the 'health professional domain', 2 items can be answered by choosing 1 of 2 options. The option associated with low therapy observance has a score of 1, while the option reflecting high therapy observance has a score of 2.
  The TAI will be completed at Visit 1 and Visit 4. The questionnaire will be made available on paper. Subjects will complete the 'patient domain' while the Investigator will complete the 'health professional domain'.

CONTACTS AND LOCATIONS:
Locations (13):
- Germany (13):
  - Thoraxklinik Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - MVZ Dachau, Dachau, Bavaria
  - Lunge im Zentrum, Erlangen, Bavaria
  - Herzzentrum des Universitätsklinikums Bonn, Bonn
  - Krankenhaus der Augustinerinnen, Cologne
  - Lungenzentrum Darmstadt, Darmstadt
  - Studienzentrum Dr. Keller, Frankfurt am Main
  - Marienkrankenhaus Kassel - Pneumologie, Kassel
  - Allgemeinmedizin Untermenzing, München
  - Lungenärzte am Rundfunkplatz, München
  - Facharztpraxis für Innere Medizin - Pneumologie - Allergologie, Oberursel
  - Lungenarztpraxis Dr. med. Maria Weber, Wiesbaden
  - Pneumologische Praxis Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun;105(6):930-8. doi: 10.1016/j.rmed.2011.01.005. Epub 2011 Mar 2. PMID 21367593
- [Background] Normansell R, Kew KM, Mathioudakis AG. Interventions to improve inhaler technique for people with asthma. Cochrane Database Syst Rev. 2017 Mar 13;3(3):CD012286. doi: 10.1002/14651858.CD012286.pub2. PMID 28288272
- [Background] O'Dwyer S, Greene G, MacHale E, Cushen B, Sulaiman I, Boland F, Bosnic-Anticevich S, Mokoka MC, Reilly RB, Taylor T, Ryder SA, Costello RW. Personalized Biofeedback on Inhaler Adherence and Technique by Community Pharmacists: A Cluster Randomized Clinical Trial. J Allergy Clin Immunol Pract. 2020 Feb;8(2):635-644. doi: 10.1016/j.jaip.2019.09.008. Epub 2019 Sep 27. PMID 31568927
- [Background] Sulaiman I, Greene G, MacHale E, Seheult J, Mokoka M, D'Arcy S, Taylor T, Murphy DM, Hunt E, Lane SJ, Diette GB, FitzGerald JM, Boland F, Sartini Bhreathnach A, Cushen B, Reilly RB, Doyle F, Costello RW. A randomised clinical trial of feedback on inhaler adherence and technique in patients with severe uncontrolled asthma. Eur Respir J. 2018 Jan 4;51(1):1701126. doi: 10.1183/13993003.01126-2017. Print 2018 Jan. PMID 29301919